CLINICAL TRIAL: NCT06377527
Title: Establishing a Tumor Registry of Patients With Mesonephric-like Adenocarcinoma (MLA)
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0945; NCI-2024-03342 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-04-16; First posted 2024-04-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mesonephric-like Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mesonephric-like Adenocarcinoma (MLA): Particpants who agree to take part in this research, information such as your demographics (including your name, date of birth, race, etc.), medical history, surgical history, family history, social history, cancer diagnosis, primary treatment, and follow up will be collected.
  Participants also have the option to agree to the use of your previously collected tumor tissue samples for future research to better understand MLA.

SUMMARY:
To develop a database of medical information about patients with MLA in an effort to increase our understanding of the characteristics of MLA, which is the rarest form of endometrial carcinoma.

DETAILED DESCRIPTION:
Primary Objectives

1. To collect data on participants characteristics, disease characterization, pathology and molecular data, treatment, and outcomes for participants with gynecologic mesonephric-like adenocarcinoma (MLA).

Secondary Objectives

1. To organize clinical information to support multifaceted queries of participant characteristics, treatment, and disease outcome data and to facilitate correlation of these characteristics with participant outcome.
2. To have a single data repository kept on a secure platform that will integrate clinical information and research findings and serve as an archive for future research.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over the age of 18.
2. Patients with a diagnosis of gynecologic mesonephric-like adenocarcinoma (MLA), mesonephric adenocarcinoma (MA), mesonephric carcinosarcoma, or mesonephric-like carcinosarcomas.
3. For patients who provide consent, they must speak and/or read English or Spanish.

Exclusion Criteria:

1. Patients with other subtypes of EACs.
2. Patients who are considered cognitively impaired. Assessment will be obtained based on their need of a Legally Authorized Representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2035-12-28 (Estimated); Study Completion 2037-12-28 (Estimated)

PRIMARY OUTCOMES:
Tumor Registry | Through study completion; an average of 1 year
  The goal of this data collection study is to develop a database (i.e. a registry/repository) of medical information about patients with MLA in an effort to increase our understanding of the characteristics of MLA, which is the rarest form of endometrial carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey How, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org